CLINICAL TRIAL: NCT00197886
Title: Dose of Norepinephrine and the Concentration of L-Lactate in the Rectum and Stomach in Patients With Septic Shock.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-7041-20
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Pressure

INTERVENTIONS:
Drug: Changing dose of norepinephrine and blood pressure

SUMMARY:
Norepinephrine is a drug used to increase blood pressure in patients with life-threatening infection. However, norepinephrine may limit the bloodflow to the gut, thereby causing relative lack of oxygen to the cells. This leads to increased formation of lactic acid.

This study examines whether increasing the dose of norepinephrine leads to higher concentrations of lactic acid in the rectum and stomach in patients with life-threatening infection.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock
* NE-dose > 0.1 microg/kg/min
* CI > 3.0 l/min/m2

Exclusion Criteria:

* Age < 18, unable to obtain informed consent from relatives
* Untreated hypertension
* Pregnancy
* Pathology in the rectum or stomach
* Limitation of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-10; Study Completion 2005-12

PRIMARY OUTCOMES:
L-lactate concentration in the rectum and stomach.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, MD,PhD, Study Chair — Dept. of Anaesthesia and Intensive Care, Herlev University Hospital, DK-2730 Herlev
Locations (1):
- Dept. of Intensive Care, Herlev University Hospital, Herlev, Denmark